CLINICAL TRIAL: NCT03725787
Title: Pressure Ulcer Incidence Cat. II+ on the CuroCell SAM® PRO Static Air Mattress: a Multicenter Cohort Study in Nursing Home Residents at Risk
Brief Title: Pressure Ulcer Incidence Cat. II+ on a Static Air Mattress: a Multicenter Cohort Study in Nursing Home Residents at Risk
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Ghent (Other)
Collaborators: Care of Sweden (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: EC/2018/0091; B670201835095 (Other: Ethics Committee UZ Gent)
Record Dates: First submitted 2018-10-25; First posted 2018-10-31 (Actual); Last update posted 2021-05-06 (Actual); Status verified 2018-10

CONDITIONS: Pressure Ulcer; Pressure Injury; Pressure Sore; Bed Sore
Keywords: Static air support surface; Support device; Elderly; Prevention
MeSH Terms: conditions — Pressure Ulcer

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CuroCell S.A.M. ® pro mattress (Experimental): Mattresses of eligible participants will be replaced by a static air pressure redistribution mattress (CuroCell S.A.M. ® Pro).
  Interventions: Device: CuroCell S.A.M. ® pro mattress

INTERVENTIONS:
Device: CuroCell S.A.M. ® pro mattress — During 30 days, participants will use the static air mattress.

SUMMARY:
Pressure Ulcers are a serious and common problem for residents admitted to long-term care facilities and community care patients. They represent a major burden to patients, carers and the Healthcare system, affecting approximately 1 in 20 community patients. International guidelines recommend the use of pressure redistribution support surfaces, systematic patient repositioning and preventive skin care to prevent pressure ulcers.

It has been acknowledged that a significant proportion of pressure ulcers are avoidable. The prevalence of pressure ulcers is 1 of the 4 common harms recorded in the UK NHS Safety Thermometer, a local improvement tool for measuring, monitoring and analyzing patient harms across a range of settings, including nursing homes, community nursing and hospitals on a monthly basis.

Static or reactive overlay mattresses are an example of a low-tech constant low-pressure support. Static air mattresses maintain a continuous low air pressure that exerts a pressure redistributing effect. Serraes and Beeckman found a pressure ulcer incidence of 5.1% in patients placed on static air support (mattress overlay, heel wedge and seat cushion) in a high risk population in a nursing home setting in Belgium.

The CuroCell SAM PRO (Care of Sweden AB) is a static air mattress overlay system used as prevent and treat pressure ulcers (up to category 3) and for pain therapy. The aim of current study is to measure pressure ulcer incidence on the CuroCell Sam PRO static air mattress in nursing home residents at risk for pressure ulcer development over a 30-day period in Belgium.

ELIGIBILITY:
Inclusion Criteria:

* At risk of pressure ulcer development based on a Braden score ≤ 17
* Bedbound or chair bound
* Aged ≥ 65

Exclusion Criteria:

* Short-stay residents (expected length of stay ≤14 days)
* End of life care
* Medical contraindication for patient repositioning/turning
* Pressure ulcer Cat. II+ present on initial evaluation

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 180 (Actual)
Dates: Start 2018-03-04 (Actual); Primary Completion 2019-02-06 (Actual); Study Completion 2020-10-06 (Actual)

PRIMARY OUTCOMES:
Pressure ulcer incidence (Cat. II+), (NPUAP classification system) | 30 days
  Development of at least 1 pressure ulcer Cat. II+ during study period, not associated with the use of medical devices

SECONDARY OUTCOMES:
Incidence rate of Cat. I pressure ulcers, (NPUAP classification system) | 30 days
  Development of at least 1 pressure ulcer Cat. I during study period, not associated with the use of medical devices
Comfort of participants (self developed questionnaire) | 30 days
  A quantitative approach to obtain insight in residents' experiences and perceptions of comfort by using a questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Dimitri Beeckman, Phd, Principal Investigator — Study Principal Investigator
Locations (8):
- Belgium (8):
  - WZC Sint-Vincentius, Deinze, Oost-Vlaanderen
  - WZC Sint-Jozef, Ghent, Oost-Vlaanderen
  - WZC Sint-Vincentius, Kaprijke, Oost-Vlaanderen
  - WZC Brugse Vaart, Mariakerke, Oost-Vlaanderen
  - Provinciaal Zorgcentrum Lemberge, Merelbeke, Oost-Vlaanderen
  - WZC Onderdale, Ursel, Oost-Vlaanderen
  - Residentie Vroonstalle, Wondelgem, Oost-Vlaanderen
  - WZC Sint-Rafaël, Liedekerke, Vlaams-Brabant

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] National Pressure Ulcer Advisory Panel, European Pressure Ulcer Advisory Panel and Pan Pacific Pressure Injury Alliance. Prevention and Treatment of Pressure Ulcers: Quick Reference Guide. Emily Haesler (Ed.). Cambridge Media: Osborne Park, Western Australia; 201.
- [Background] Levy A, Kopplin K; BS; Gefen A. Computer simulations of efficacy of air-cell-based cushions in protecting against reoccurrence of pressure ulcers. J Rehabil Res Dev. 2014;51(8):1297-319. doi: 10.1682/JRRD.2014.02.0048. PMID 25625315
- [Background] Brown S, Smith IL, Brown JM, Hulme C, McGinnis E, Stubbs N, Nelson EA, Muir D, Rutherford C, Walker K, Henderson V, Wilson L, Gilberts R, Collier H, Fernandez C, Hartley S, Bhogal M, Coleman S, Nixon JE. Pressure RElieving Support SUrfaces: a Randomised Evaluation 2 (PRESSURE 2): study protocol for a randomised controlled trial. Trials. 2016 Dec 20;17(1):604. doi: 10.1186/s13063-016-1703-8. PMID 27993145
- See also: Website of the research group — https://www.skintghent.be/en